CLINICAL TRIAL: NCT01360996
Title: Positive Clinical and Hormonal Effects of Ethinylestradiol Combined With Drospirenone (EE/DRSP) in Women With Polycystic Ovary Syndrome (PCOS): Impact of Body Weight and Relevance to Hyperandrogenism
Brief Title: Low Dose OC Therapy in Women With Polycystic Ovary Syndrome (PCOS): Impact of BMI on Hyperandrogenism
Acronym: BEYAZ-PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Principal Investigator, Karen Elkind-Hirsch, Scientific Director of Research, Woman's
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP 11-003
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — beyaz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3 mg DRSP/20 μg EE--normal weight (Experimental): Folate-boosted 3 mg DRSP/20 μg EE-24/4 oral contraceptive
  Normal weight -BMI 18-24.9 kg/ m2
  Interventions: Drug: 3 mg DRSP/20 μg EE
- 3 mg DRSP/20 μg EE- Overweight (Experimental): Folate-boosted 3 mg DRSP/20 μg EE-24/4 oral contraceptive
  BMI 25-29.9 kg/ m2
  Interventions: Drug: 3 mg DRSP/20 μg EE
- 3 mg DRSP/20 μg EE- Grade 1 obese (Experimental): Folate-boosted 3 mg DRSP/20 μg EE-24/4 oral contraceptive
  BMI 30-34.9 kg/ m2
  Interventions: Drug: 3 mg DRSP/20 μg EE

INTERVENTIONS:
Drug: 3 mg DRSP/20 μg EE — 1 pill daily-24 days of drospirenone 3 mg (3 mg DRSP)/ethinyl estradiol 20 μg (20 μg EE)/levomefolate calcium 0.451 mg (folate) -followed by 4 days of levomefolate calcium 0.451 mg (folate)only
  Other Names: folate-boosted 3 mg DRSP/20 μg EE-24/4 oral contraceptive; BeYaz

SUMMARY:
The classic description of polycystic ovary syndrome (PCOS) is that it is a disorder characterized by menstrual irregularity, chronic anovulation, androgen excess, and abnormal gonadotropin secretion. Use of combined oral contraceptives (OCs) in women with PCOS effectively reduces circulating androgens. Although OCs are the most common and one of the oldest symptomatic treatment modalities for androgenic skin symptoms and for irregular menstrual cycles caused by hyperandrogenism, the data concerning the effect of treatment of PCOS women with different body mass index (BMI) are limited. This study is being done to compare the hormone and metabolic changes after treatment with low-dose oral birth control regimen of DRSP 3 mg/EE 0.02mg/levomefolate calcium 0.451 mg (Beyaz™) in women with PCOS with different body weights.

DETAILED DESCRIPTION:
Clinically, polycystic ovary syndrome (PCOS) is a heterogeneous disorder of functional androgen excess and the features of PCOS can run through a spectrum of severity. The optimal modality for long-term treatment of PCOS should positively influence androgen synthesis, sex hormone binding globulin (SHBG) production, insulin sensitivity, the lipid profile, and clinical symptoms including hirsutism and irregular menstrual cycles. Combined oral contraceptives have been a key component of the chronic treatment of women with PCOS; improving androgen excess and regulating menstrual cycles. The effect of OCs on ovarian folliculogenesis significantly decreases androgen production. This mechanism was confirmed in both healthy women and women with PCOS. In obese patients with PCOS, it is likely that the suppression of androgen production is not as significant. It is thus possible to hypothesize that the effects of OCs in PCOS could be dependent on body weight and what is needed is a head-to-head comparison. The aim of this study is to compare the effect of 6 months of a low-dose oral contraceptive regimen of 24/4 DRSP 3 mg/EE 0.02mg/levomefolate calcium 0.451 mg on androgen profiles, cardiometabolic measures, B-vitamin status, and menstrual cycle regulation in three groups, normal (BMI 18-24.9 kg/ m2) overweight (BMI 25-29.9 kg/ m2) and obese (BMI 30-35 kg/ m2) women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* •Adult female-16 years to 35 years of age who have been diagnosed with PCOS desiring contraception

  * Actual BMI >18 to <35kg/ m2
  * Written consent for participation in the study
  * Patient completed lactation

Exclusion Criteria:

* Metabolic abnormalities requiring pharmacological intervention (except controlled thyroid disease)

  * Uncontrolled hypertension
  * Cancer or history of hormone-dependent cancer
  * History of cholestasis
  * Presence of contradictions for OC administration
  * Personal history of cardiovascular events.
  * Use of drugs known to exacerbate glucose tolerance.
  * No prescription or over-the-counter weight-loss drugs
  * Diabetes
  * Use of medications that affect blood pressure or lipid profile
  * Smoking in past 6 months
  * Known thrombogenic mutations (e.g. Factor V Leiden)
  * Current or history of deep venous thrombosis/pulmonary embolism
  * Major surgery with prolonged immobilization
  * Injectable hormonal contraceptive use within 6 months
  * Use of hormonal (e.g., oral contraceptive [OC] pill) or insulin-sensitizing medication unless willing to cease medications for 3 months before study measurements

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2011-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Elkind-Hirsch, M.Sc.,Ph.D., Principal Investigator — Woman's Hospital, Louisiana; Martha Paterson, M.D., Principal Investigator — Woman's Hospital Metabolic Health Clinic
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This clinical trial was conducted from January 2012 to December 2014 Healthy, premenopausal women (n=64) with polycystic ovary syndrome (PCOS), aged between 16 and 35 years inclusive with a baseline body mass index (BMI) of >18 to <35kg/ m2, recruited from Woman's Metabolic Health clinic and Woman's Hospital gynecology clinics were enrolled
Pre-assignment Details: Diabetic subjects, smokers, injectable hormonal contraceptive use within 6 months, or those taking sex hormones, carbohydrate metabolism, lipid-lowering and/or anti-obesity drugs within 3 months of the study were excluded
Groups:
- 3 mg DRSP/20 μg EE--normal Weight: Folate-boosted 3 mg DRSP/20 μg EE-24/4 oral contraceptive
  Normal weight -BMI 18-24.9 kg/ m2
  3 mg DRSP/20 μg EE: 1 pill daily-24 days of drospirenone 3 mg (3 mg DRSP)/ethinyl estradiol 20 μg (20 μg EE)/levomefolate calcium 0.451 mg (folate) -followed by 4 days of levomefolate calcium 0.451 mg (folate)only
- 3 mg DRSP/20 μg EE- Overweight: Folate-boosted 3 mg DRSP/20 μg EE-24/4 oral contraceptive
  BMI 25-29.9 kg/ m2
  3 mg DRSP/20 μg EE: 1 pill daily-24 days of drospirenone 3 mg (3 mg DRSP)/ethinyl estradiol 20 μg (20 μg EE)/levomefolate calcium 0.451 mg (folate) -followed by 4 days of levomefolate calcium 0.451 mg (folate)only
- 3 mg DRSP/20 μg EE- Grade 1 Obese: Folate-boosted 3 mg DRSP/20 μg EE-24/4 oral contraceptive
  BMI 30-34.9 kg/ m2
  3 mg DRSP/20 μg EE: 1 pill daily-24 days of drospirenone 3 mg (3 mg DRSP)/ethinyl estradiol 20 μg (20 μg EE)/levomefolate calcium 0.451 mg (folate) -followed by 4 days of levomefolate calcium 0.451 mg (folate)only
Period: Overall Study
Arm/Group | 3 mg DRSP/20 μg EE--normal Weight | 3 mg DRSP/20 μg EE- Overweight | 3 mg DRSP/20 μg EE- Grade 1 Obese
Started | 20 | 21 | 23
Completed | 14 | 18 | 21
Not Completed | 6 | 3 | 2
Not completed — Withdrawal by Subject | 4 | 3 | 2
Not completed — Noncompliant | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: oligomenorrhea and biochemical hyperandrogenism (total T >1.38 nmol/l or free androgen index [FAI] >3.87) and exclusion of other etiologies (non-classic congenital adrenal hyperplasia, androgen-secreting tumors, hyperprolactinemia, Cushing syndrome, thyroid dysfunction and primary ovarian insufficiency
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mg DRSP/20 μg EE--normal Weight | 3 mg DRSP/20 μg EE- Overweight | 3 mg DRSP/20 μg EE- Grade 1 Obese | Total
Number analyzed (Participants) | 20 | 21 | 23 | 64
Age, Categorical [Count of Participants; unit: Participants] — Healthy, premenopausal women (n=64) with polycystic ovary syndrome (PCOS), aged between 16 and 35 years inclusive with a body mass index (BMI) of >18 to <35kg/ m2,
  Participants
    <=18 years | 3 | 2 | 4 | 9
    Between 18 and 65 years | 17 | 19 | 19 | 55
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 23 | 64
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 23 | 64

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Assessment of Hyperandrogenism
Description: The primary outcome measure is post-treatment Free Androgen Index(FAI) which is expressed in units.
  FAI is calculated by taking the testosterone concentration (in nmol/l) and dividing by concentration of sex hormone binding globulin (SHBG in nmol/L)and multiplying by 100
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Non-Obese: There was no significant difference on any variables between normal and overweight at baseline so groups were combined into non-obese
  Folate-boosted 3 mg DRSP/20 ug EE-24/4 oral contraceptive
  BMI 18-29.9 kg/m2
- Obese: Folate-boosted 3 mg DRSP/20 ug EE-24/4 oral contraceptive
  BMI 30-34.9 kg/m2 (obese grade 10
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 32 | 21
Index | 0.7 (0.5) | 0.7 (0.45)
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Test type: Superiority or Other; p < .0001, ANOVA

2. Secondary Outcome: Cardiometabolic Measures
Description: Values represent blood pressure at 24 weeks.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 32 | 21
mmHg | 120 (13) | 125 (9)
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Test type: Superiority or Other; p > 0.05, ANOVA

3. Secondary Outcome: Post Therapy BMI.
Description: Post-treatment body mass index at 24 weeks
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 32 | 21
kg/m2 | 24.6 (3.9) | 32.7 (2.7)
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Test type: Superiority or Other; p > 0.05, ANOVA

4. Secondary Outcome: Biochemical Indicator of B-vitamin Status
Description: Post-treatment in folate concentrations after 24 weeks of treatment
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Folate in nmol/l
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 32 | 21
Folate in nmol/l | 65.8 (20.4) | 60.8 (20.6)
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Test type: Superiority or Other; p < 0.001, ANOVA

5. Secondary Outcome: Menstrual Cycle Regularity
Description: Post treatment menstrual frequency over 24 weeks normalized to number of menses per year ..
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: number of cycles annually
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 32 | 21
number of cycles annually | 11.3 (1.7) | 11 (1.4)
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Test type: Superiority or Other; p < 0.0001, McNemar

6. Secondary Outcome: Adrenal Androgen DHEAS
Description: Post-treatment levels of adrenal androgen DHEAS
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 32 | 21
micromol/L | 4.9 (2.2) | 4.3 (2.3)
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Test type: Superiority or Other; p < 0.001, ANOVA

7. Secondary Outcome: Oral Disposition Index
Description: Post-treatment insulin secretion-sensitivity index (ISSI) calculated from the oral glucose tolerance test (OGTT). A higher value indicate improved carbohydrate metabolism
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: calculated index
Arm/Group | Non-Obese | Obese
Number analyzed (Participants) | 32 | 21
calculated index | 732 (420) | 272 (226)
Statistical Analysis 1: Comparison: Non-Obese vs Obese; Test type: Superiority or Other; p < 0.04, ANOVA

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 3 mg DRSP/20 μg EE--normal Weight | 3 mg DRSP/20 μg EE- Overweight | 3 mg DRSP/20 μg EE- Grade 1 Obese
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/23

LIMITATIONS AND CAVEATS:
Limitations include evaluation after 24 weeks in a limited number of patients, The time may be too short and sample size too small to measure differences between normal and overweight PCOS women and the use of indirect measures of insulin action.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes